CLINICAL TRIAL: NCT07054853
Title: Effect of Induced Rotator Cuff Muscles Fatigue on Hand Grip Strength in Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Noura Karam Abdou Mohammed Ismaiel (Other)
Collaborators: Cairo University (Other); Misr University for Science and Technology (Other)
Responsible Party: Sponsor-Investigator, Noura Karam Abdou Mohammed Ismaiel, Teaching Assistant, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/005798
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy Individuals
Keywords: muscle fatigue; neuromuscular performance; isokinetic biodex; hand grip strength; rotator cuff muscles

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group males and females
  Interventions: Device: Induced rotator cuff fatigue by isokinetic biodex

INTERVENTIONS:
Device: Induced rotator cuff fatigue by isokinetic biodex — Each subject will undergo two separate fatigue protocols from distinct shoulder abduction angles (30° and 90°), referred to as Protocol A and Protocol B, respectively.
  Fatigue will be induced using the Biodex System 4 Pro Isokinetic .Participants will be seated with the tested arm positioned at the designated shoulder abduction angle and elbow flexed at 90°. The arm will be secured using a shoulder adapter to ensure standardized positioning. Hand Grip strength will be assessed using a Jamar Plus+ Digital. Participants will perform three maximal grip trials, each lasting 3 seconds, with verbal encouragement provided. The average of the three trials will be used as the maximum voluntary contraction

SUMMARY:
This observational study aims to investigate the effect of induced rotator cuff muscles fatigue on hand grip strength in adults

DETAILED DESCRIPTION:
This study is set to take place at the Isokinetic Biodex Laboratory, Faculty of Physical Therapy at Misr University for Science and Technology (MUST). The goal is to explore how fatigue in the rotator cuff muscles affects hand grip strength in healthy adults.

The study will involve 30 healthy male and female participants, aged between 18 and 30 years, all recruited from the university. To ensure the reliability of the results, participants must meet specific inclusion criteria: they should have no recent history of shoulder or back pain, no spinal deformities, and a body mass index within the normal range. Individuals with any upper limb disorders, recent surgeries, or neurological issues will be excluded.

The experimental protocol is carefully structured and will be conducted using two key tools. The first is the Biodex System 4 Pro, an isokinetic dynamometer renowned for its accuracy in measuring muscle performance and fatigue. The second is the Jamar Plus+ Digital, a gold-standard device for measuring grip strength, known for its reliability and ease of use.

Participants will attend two fatigue sessions apart to prevent carryover effects. Each session will involve a fatigue protocol by isokinetic biodex system targeting the shoulder's internal and external rotators at two different abduction angles: 30° (Protocol A) and 90° (Protocol B).

Grip strength will be assessed both before and after each fatigue session using the Jamar plus+ Digital. Participants will sit with their arms and legs positioned for standardized testing, and each will complete three maximal grip trials. The average of these attempts will be recorded, with verbal encouragement provided to ensure maximal effort.

Through this structured investigation, the study aims to shed light on how rotator cuff fatigue influences hand grip strength-an insight that could have practical implications for injury prevention, rehabilitation strategies, and performance optimization in both clinical and athletic settings.

ELIGIBILITY:
Inclusion Criteria:

* Both male and females (18-30) years
* No complaints of existing shoulder pathology/pain in at least one shoulder within the last 6 months, no back pain, no history of shoulder/thoracic spine surgery, and no spinal deformities
* Body mass index between (18.5:24.99) Kg/ m2

Exclusion Criteria:

* Shoulder complaints in the past 6 months such as shoulder dislocation rotator cuff tear, shoulder surgery, and shoulder rehabilitation or other upper limb forms of disability
* Subjects who had wrist pain, a joint injury, undergone surgery, or neuromuscular dysfunction were excluded from the study
* Individuals who suffered an injury or underwent a surgical procedure in the last six months that could affect hand functions or senses

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy Individuals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Hand Grip Strength | 3 months
  Maximum Voluntary Contraction

CONTACTS AND LOCATIONS:
Locations (1):
- Misr University for Science and Technology, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No